CLINICAL TRIAL: NCT00755456
Title: Phase 2 Study of the Effect of a Peritoneal Dialysis Solution Containing Glucose (1.5%) and L-carnitine (0.1%) on Insulin Sensitivity in Patients on Continuous Ambulatory Peritoneal Dialysis
Brief Title: Effect of an L-carnitine-containing Peritoneal Dialysis (PD) Solution on Insulin Sensitivity in Patients on Continuous Ambulatory Peritoneal Dialysis (CAPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Iperboreal Pharma Srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IP-002-05
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2013-03

CONDITIONS: End Stage Renal Disease; Insulin Resistance
Keywords: Peritoneal dialysis; L-carnitine; Insulin resistance; Glucose homeostasis; Dyslipidemia
MeSH Terms: conditions — Kidney Failure, Chronic; Insulin Resistance; Dyslipidemias | interventions — Carnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucose solution (Active Comparator)
  Interventions: Drug: PD solution containing glucose
- Glucose and L-carnitine solution (Experimental)
  Interventions: Drug: PD solution containing glucose and L-carnitine

INTERVENTIONS:
Drug: PD solution containing glucose — Instillation of PD solutions containing Glucose (1.5 or 2.5%, w/v) for the diurnal exchanges, and 1 PD solution containing icodextrin (7.5 w/v) for nocturnal exchange. PD solutions are instilled for 120 days.
  Other Names: Dianeal (Baxter)
  Arms: Glucose solution
Drug: PD solution containing glucose and L-carnitine — Instillation of PD solutions containing Glucose (1.5 or 2.5%, w/v) and L-carnitine (0.1%, w/v) for the diurnal exchanges, and 1 PD solution containing icodextrin (7.5 w/v) for nocturnal exchanges. PD solutions are instilled for 120 days.
  Arms: Glucose and L-carnitine solution

SUMMARY:
The current study is initiated in order to assess the impact of a PD solution containing L-carnitine on insulin sensitivity measured by a hyperinsulinemic euglycemic clamp.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Have a diagnosis of ESRD and have been on Continuous Ambulatory Peritoneal Dialysis (CAPD) for at least 3 months
3. Be in a stable clinical condition during the four weeks immediately prior to Screening Period as demonstrated by medical history, physical examination and laboratory testing
4. Have a blood hemoglobin concentration above 8,5 g/100ml (data will be verified with Investigators)
5. Have not experienced peritonitis episodes in the last 3 months
6. Be treated with Extraneal (nocturnal exchange bag solution) for at least 1 month
7. Be treated with 3 diurnal exchange bag solutions (1.5% or 2.5% glucose) and one nocturnal exchange bag solution (Extraneal)
8. Have Kt/V urea measurement > 1.7 per week in a previous test performed within 6 months that should be confirmed at Baseline Visit
9. Have a minimum weekly creatinine clearance of 45 litres in a previous test performed within 6 months that should be confirmed at Baseline Visit
10. Have a D/P Creatinine ratio at Peritoneal Equilibration Test (PET) between 0.50 and 0.81 in a previous test performed within 6 months that should be confirmed at Baseline Visit
11. Have a D/P Glucose ratio at Peritoneal Equilibration Test (PET) between 0.26 and 0.49 in a previous test performed within 6 months that should be confirmed at Baseline Visit
12. Be treated by the participating clinical Investigator for a period of at least three months
13. Have understood and signed the Informed Consent Form.

Exclusion Criteria:

1. Have a history of drug or alcohol abuse in the six months prior to entering the protocol
2. Be in treatment with androgens
3. Have Diabetes Mellitus (as defined by the American Diabetes Society, objectively documented by a fasting plasma glucose and HbA1c determinations)
4. Have clinically significant abnormal liver function test (SGOT, SGPT, and gamma-GT > 2 times the upper normal limit)
5. Have acute infectious conditions (i.e.: pulmonary infection, acute hepatitis, high or low urinary tract infections, renal parenchymal infection, pericarditis, etc)
6. Have a history of congestive heart failure and clinically significant arrhythmia
7. Have an history of epilepsy or any NCS disease
8. Have malignancy within the past 5 years, including lymphoproliferative disorders
9. Have any medical condition that, in the judgment of the Investigator, would jeopardize the patient's safety following exposure to study drug, particularly if patient's life expectancy is less than 1 year
10. Have a history of L-Carnitine therapy or use in the month prior to entering the protocol
11. Have used any investigational drug in the 3 months prior to entering the protocol
12. Be in pregnancy, lactation, fertility age without protection against pregnancy by adequate contraceptive means

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of L-Carnitine containing PD solution on insulin sensitivity evaluated by euglycemic hyperinsulinemic clamp | time 0, 4 months

SECONDARY OUTCOMES:
To assess the efficacy of L-Carnitine containing PD solution on plasma lipids and lipoprotein profile | -2 weeks, time 0, 1 month, 2 months, 3 months, 4 months
To assess the efficacy of L-Carnitine containing PD solution on hematological parameters (hemoglobin and EPO requirements) | -2 weeks, time 0, 2 months, 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Mario Bonomini, MD, Principal Investigator — G. d'Annunzio University; Arduino Arduini, MD, Study Director — Iperboreal Pharma Srl
Locations (12):
- Italy (12):
  - Renal and Dialysis, Bari Policlinic Hospital, Bari
  - Renal, Dialysis and Transplant Unit, University of Bari, Bari
  - Division of Nephrology, University of "G. d'Annunzio", Chieti
  - Nephrologyand Dialysis Unit, Desio Hospital, Desio
  - Nephrology and Dialysis Unit, "Maria SS dello Splendore" Hospital, Giulianova
  - Nephrology and Dialysis Unit, "Renzetti" Hospital, Lanciano
  - Division of Nephrology and Dialysis, Ospedale Policlinico Maggiore, Milan
  - Nephrology and Dialysis Unit, "G. Bernabeo" Hospital, Ortona
  - Renal Unit, Policlinico MultiMedica, Sesto San Giovanni
  - Nephrology and Dialysis Unit, "SS Annunziata" Hospital, Sulmona
  - Division of Nephrology and Dialysis, "Mazzini" Hospital, Teramo
  - Nephrology and Dialysis Unit, "San Pio da Pietrelcina" Hospital, Vasto

REFERENCES:
- [Result] Bonomini M, Di Liberato L, Del Rosso G, Stingone A, Marinangeli G, Consoli A, Bertoli S, De Vecchi A, Bosi E, Russo R, Corciulo R, Gesualdo L, Giorgino F, Cerasoli P, Di Castelnuovo A, Monaco MP, Shockley T, Rossi C, Arduini A. Effect of an L-carnitine-containing peritoneal dialysate on insulin sensitivity in patients treated with CAPD: a 4-month, prospective, multicenter randomized trial. Am J Kidney Dis. 2013 Nov;62(5):929-38. doi: 10.1053/j.ajkd.2013.04.007. Epub 2013 May 29. PMID 23725973
- [Derived] Nishioka N, Luo Y, Taniguchi T, Ohnishi T, Kimachi M, Ng RC, Watanabe N. Carnitine supplements for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013601. doi: 10.1002/14651858.CD013601.pub2. PMID 36472884